CLINICAL TRIAL: NCT06371755
Title: REMS Versus DXA for Bone Mineral Density (BMD) Evaluation
Brief Title: Bone Evaluation by Ultrasound Radiofrequency Echographic Multi Spectrometry (REMS) vs Dual X-ray Absorptiometry (DXA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paola Pisani (Industry)
Collaborators: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor-Investigator, Paola Pisani, Clinical Director, Echolight S.p.A.
Organization: Echolight S.p.A. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ULTRADXA
Record Dates: First submitted 2024-03-08; First posted 2024-04-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis Diagnosis
Keywords: REMS,; Femur; Spine; DXA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Execution of additional diagnostic examination (Other): The proposed study is defined as interventional because it introduces an ultrasound examination in the standard clinical routine. The diagnostic approach does not vary during the study and the prescription of any therapeutic treatment is performed on the basis of the conventional DXA diagnosis. This ultrasound examination does not involve additional risks for the patient with the benefit of not using ionizing radiation; it lasts only few minutes and can be performed without moving the patient from the same bed on which he is already positioned for DXA examination.
  Interventions: Device: Ultrasound examination with REMS technology

INTERVENTIONS:
Device: Ultrasound examination with REMS technology — The proposed study is defined as interventional because it introduces an ultrasound examination in the standard clinical routine. The diagnostic approach does not vary during the study and the prescription of any therapeutic treatment is performed on the basis of the conventional DXA diagnosis. This ultrasound examination does not involve additional risks for the patient with the benefit of not using ionizing radiation; it lasts only few minutes and can be performed without moving the patient from the same bed on which he is already positioned for DXA examination.

SUMMARY:
Bone Density Evaluation by means of the Ultrasound Technology Named Radiofrequency Echographic Multi Spectrometry (REMS) in Comparison With DXA Technique.

Clinical Center involved in the study:IRCCS Orthopedic institute Galeazzi - Sant'Ambrogio The clinical study will evaluate the intra- and inter-operator repeatability of the REMS,(Radiofrequency Echographic Multi Spectrometry) ultrasound diagnostic technology implemented in the EchoStation device (Echolight Spa, Lecce) and the diagnostic accuracy in comparison with DXA (used as standard reference).

DETAILED DESCRIPTION:
The study protocol was approved by the Ethics Review Boards of the Galeazzi Hospital in Milan (Comitato Etico San Raffaele, Milano, Italy). According to the protocol, only women will be enrolled because they are the vast majority of subjects usually tested for BMD using DXA. Women who voluntarily entered the study, will provide written informed consent and authorization for anonymized data publication.

To determine the short-term intra-operator precision and inter-operator repeatability of radiofrequency echographic multi-spectrometry (REMS) at the lumbar spine (LS) and proximal femur (FEM). All patients will undergo an ultrasound scan of the LS and FEM. Both precision and repeatability, expressed as root-mean-square coefficient of variation (RMS-CV) and least significant change (LSC) will be evaluated using data from two consecutive REMS acquisitions by the same operator or two different operators, respectively. The precision will be also assessed in the cohort stratified according to BMI classification.

To evaluate the comparison between REMS and DXA diagnostic results, spinal DXA reports were processed separately from femoral ones. According to spinal DXA reports, each patient was classified as osteoporotic^ if lumbar T-score≤ -2.5 and as non-osteoporotic if lumbar T-score > -2.5. An independent classification employing the same threshold was adopted on the basis of femoral neck T-score values obtained from femoral DXA reports. In both cases the non-osteoporotic patients were further classified as osteopenic if -2.5 < T-score < -1.0 or healthy^ if T-score≥ -1.0.

The whole classification process was independently repeated on the basis of the corresponding lumbar and femoral neck T-score values obtained from REMS scans.

Diagnostic accuracy of the REMS approach was then assessed by assuming DXA outputs as the standard reference. The diagnostic concordance between the two methods was assessed, by calculating the percentage of patients being classified in the same diagnostic category (osteoporotic, osteopenic, or healthy) by both DXA and REMS together with the degree of correlation between DXA and REMS T-score values.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for lumbar and/or femoral DXA examination,
* female sex,
* age range 30-80 years (for repeatability study), age range 50-70 years (for accuracy study),
* absence of severe obesity (BMI < 40 kg/m2),
* absence of severe walking difficulties,
* cognitive underwriting of informed consent.

Exclusion Criteria:

* Male sex,
* severe walking difficulties,
* age below 30 years or over 80 years,
* severe obesity (BMI > 40 kg/m2),
* declared pregnancy.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Women were included in the study since female population undergoes densitometric examinations more frequently that the male one.
Enrollment: 296 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. REMS Technology intra - and inter-operator repeatability Evaluation. | up to 3 months
  The Root Mean Square - Coefficient of Variation (CV-RMS) parameter has been measured in order to calculate REMS intra- and inter-operator repeatability.

SECONDARY OUTCOMES:
1. Evaluation of the accuracy of the REMS Technology in comparison with the conventional DXA technique. | through study completion, an average of 1 year
  Evaluation of the diagnostic agreement between the two used diagnostic techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Luca M. Sconfienza, Professor, Principal Investigator — IRCCS
Locations (1):
- I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No